CLINICAL TRIAL: NCT06509750
Title: The Postprandial Effects of a Carob-containing Meal
Acronym: ACM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C. Kaliora, Professor, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ACM-147
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal_1 (Experimental): Bread, butter and carob-beverage
  Interventions: Other: Carob-meal
- Meal_2 (Experimental): bread, butter and beverage with sugar (orange beverage)
  Interventions: Other: Non-carob-meal

INTERVENTIONS:
Other: Carob-meal — A meal with carob-beverage
  Arms: Meal_1
Other: Non-carob-meal — A meal with orange-beverage
  Arms: Meal_2

SUMMARY:
In an era where malnutrition and unhealthy eating patterns are salient contributors to global health deterioration, the urge for better access to nutritious alimentation is striking. Native to the Mediterranean region, the carob tree holds significant promise in this regard. With its rich nutritional profile, containing high levels of dietary fiber, polyphenols, and essential minerals, carob has been increasingly exploited by the food industry. Carob flour, derived from the pod after seed removal, is widely used as a cocoa substitute. The carob tree's fruit comprises 10% seeds and 90% pulp, containing numerous bioactive components such as dietary fiber, cyclitols, phenolic compounds, amino acids, and minerals. These components have been associated with beneficial effects on the gastrointestinal system and glucose absorption, with small-scale clinical studies indicating a hypolipidemic effect in patients with hypolipidemia. Nevertheless, comprehensive data from randomized controlled trials on the biological actions of carob remain restricted. This study explores the postprandial effects of incorporating carob into a Western-style meal, focusing on regulating glucose, insulin, and appetite hormones. The hypothesis is that a carob-enriched breakfast meal could positively influence satiety and appetite regulation, potentially offering a nutritious and sustainable dietary option for improving metabolic health. The high fiber and polyphenol content in carob are expected to modulate these postprandial responses, contributing to a better understanding of carob's role in dietary interventions. This study supports international initiatives to combat malnutrition and encourage a healthy diet, especially in light of the growing world population and the requirement for sustainable food supplies. By investigating the impact of carob on postprandial metabolic responses, this study seeks to contribute valuable insights into its potential benefits as part of a healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* healthy male adults
* normal weight

Exclusion Criteria:

high body fat mass Type 1 Diabetes, cardiovascular diseases, hypertension thyroid disorder, liver disease, kidney disease gastrointestinal disease mental illness use of nutraceutical supplements or natural products for weight loss dietitians/nutritionists

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Plasma ghrelin levels | 3 hours
  Plasma ghrelin levels in the two groups for the comparison of objective satiety between treatments.
Changes in visual analogue scale | 3 hours
  Changes in visual analogue scale for the comparison of subjective satiety between the two groups. Values range 0-10, the higher the value the higher satiety

CONTACTS AND LOCATIONS:
Locations (1):
- Andriana Kaliora, Athens, Greece